CLINICAL TRIAL: NCT02478424
Title: Extended Use of Cannabidiol for the Prevention of Graft-versus-host Disease After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Extended Use of Cannabidiol for the Prevention of Graft-versus-host-disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMC-0208-14
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cannabidiol; Cyclosporine; Methotrexate

ARMS (1):
- Cannabidiol arm (Experimental): Patients undergoing an allogeneic hematopoietic cell transplantation will be given standard GVHD prophylaxis comprising cyclosporine and a short course of methotrexate plus CBD 150 mg BID starting 7 days before transplantation until day 100.
  Interventions: Drug: Cannabidiol; Drug: cyclosporine; Drug: Methotrexate

INTERVENTIONS:
Drug: Cannabidiol — Patients will receive standard GVHD prophylaxis consisting of cyclosporine A twice daily starting on day -1 with target trough levels of 200-400 ng/mL and a short course of methotrexate (15 mg/ m2 on day 1 and 10 mg/ m2 on days days 3 and 6). Patients transplanted from unrelated donors will receive ATG Fresenius at a low dose of 5 mg/kg on days -3 to -1.
  Patients will be given oral CBD 150 mg BID starting 7 days before transplantation until day 100.
  Other Names: CBD
Drug: cyclosporine
Drug: Methotrexate

SUMMARY:
Cannabidiol (CBD), a non-psychotropic ingredient of Cannabis sativa possesses potent anti-inflammatory and immunosuppressive properties. In a recent prospective phase II study (NCT01385124) 48 consecutive adult patients undergoing allogeneic hematopoietic cell transplantation were given CBD 300 mg/day starting 7 days before transplantation until day 30, on top of standard GVHD prophylaxis consisting of cyclosporine and a short course of methotrexate. There were no grade 3-4 toxicities attributed to CBD. None of the patients developed acute GVHD while consuming CBD. With a median follow-up of 16 months, the cumulative incidence rates of grade 2-4 and grade 3-4 acute GVHD by day 100 were 12.1% and 5%, respectively. Compared to 101 historical control subjects given standard GVHD prophylaxis, the hazard ratio of developing grade 2-4 acute GVHD among subjects treated with CBD plus standard GVHD prophylaxis was 0.3 (p=0.0002). Among patients surviving more than 100 days, the cumulative incidence of moderate-to-severe chronic GVHD at 12 and 18 months were 20% and 33%, respectively.

The aim of this study is to explore the safety and efficacy of extended use of CBD until day 100 in the prevention of acute and chronic GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Acute leukemia in complete remission
2. Myeloablative conditioning
3. Matched or one antigen or allele mismatched sibling or unrelated donor

Exclusion Criteria:

1. History of psychosis
2. Bronchial asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2-4 and grade 3-4 acute GVHD by day 100 | 100 days
grade 3-4 adverse effects attributed to CBD consumption | 180 days
Incidence of overall chronic GVHD and moderate to severe chronic GVHD by 12 months | 12 months
Incidence of late onset acute GVHD | 12 months

SECONDARY OUTCOMES:
Non relapse mortality | 12 months
Relapse rate | 12 months
Overall survival | 12 months
Adherence to study protocol | Until day 100
  Percentage of doses actually taken as reported by patients
Disease free and immunosuppression free survival by 12 months | 12 months